CLINICAL TRIAL: NCT03658798
Title: Testing the Efficacy of Garment-embedded Electrodes for Functional Electrical Stimulation: Training of Individuals With Upper-limb Paralysis.
Brief Title: Grasping Rehabilitation With Functional Electrical Stimulation Garment
Acronym: GarmentGrasp
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funds have not been received
Sponsor: Milos Popovic (Other)
Responsible Party: Sponsor-Investigator, Milos Popovic, Research Director, Toronto Rehabilitation Institute
Organization: Toronto Rehabilitation Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-6348
Record Dates: First submitted 2018-06-12; First posted 2018-09-05 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Stroke; Spinal Cord Injuries
Keywords: Functional Electrical Stimulation; Neuroprosthesis; Rehabilitation
MeSH Terms: conditions — Stroke; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Participant will be compared to themselves in a "pre-post" analysis
Masking Description: No masking of the intervention to participant or assessor because there is only 1 arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FES-Garment (Experimental): All participants will take part in 40 sessions of 1 hour of Functional Electrical Stimulation
  Interventions: Procedure: Functional Electrical Stimulation

INTERVENTIONS:
Procedure: Functional Electrical Stimulation — Study participants will receive 40 sessions of intervention, 3 to 5 times a week over 2 to 3 months. Each session will be one hour in duration and participant will receive functional electrical stimulation therapy with their customized shirt. During therapy participants will be expected to carry out functional movements with assistance from the FES Garment.Participants will be expected to don, activate, and doff the garment as independently as possible. The exercises conducted will be defined by the investigator based on the functional status of the participant and eventual progress.

SUMMARY:
This study tests the feasibility, safety and efficacy of garments embedding conductive electrodes (FES-shirt) for the independent delivery of functional electrical stimulation (FES). 12 people with SCI and 12 people with stroke who have some degree of arm paralysis will receive 40 hours of FES with these FES-shirt. The ability to use the FES-shirts and the improvement in function while receiving FES will indicate the immediate benefits. Their functional capabilities will be measured before and after 40 FES sessions to evaluate the carry-over effects.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) and stroke can result in paralysis of arm and hand muscles preventing people from being able to use them in day to day activities, which can greatly impact quality of life. Functional electrical stimulation (FES) can activate the paralyzed muscles by sending a low energy electrical current through the skin. FES has been shown to improve the ability to control muscles in previous studies.In current simulators individual adhesive gel electrodes are positioned on the appropriate muscles to produce functional movements.This is time consuming and requires a therapist to guide electrode placement,besides the cables interfere with the individuals ability to perform functional movements with the FES.To approach this issue, we designed prototype shirts embedding all the necessary electrodes and wires to stimulate muscles around the hand, elbow and shoulder.

24 individuals with difficulty performing routine day to day activities with their upper extremities will be recruited to the study: 12 people with SCI and 12 people with stroke. Each participant will receive a custom designed FES shirt made based on individual participant body measurements and optimal electrode positions identified with standard gel electrodes.Study participants will receive 40 sessions of intervention, 3 to 5 times a week over 2 to 3 months. Each session will be one hour in duration and participant will receive functional electrical stimulation therapy through this customized shirt. They will have to don, activate, and doff the garment as independently as possible. The exercises conducted will be defined by the investigator based on the functional status of the participant and eventual progress.

Participants will be evaluated before and after the intervention using functional tests and questionnaires Participants will be invited to give their opinions on the shirt so that the researchers can improve its features.

ELIGIBILITY:
Inclusion Criteria:

* Complete and Incomplete C4-C7 SCI or brain vascular stroke (hemorrhagic or ischemic)
* Upper-limb paralysis to the extent that it interferes with the participants ability to perform activities of daily living independently.
* More than 6 months post injury at the time of recruitment and should have been discharged from initial post-acute rehabilitation
* Able to communicate verbally and read in English

Exclusion Criteria:

* Implanted electronic devices such as: defibrillator, stimulator, insulin pump, baclofen pump, pace maker
* Contracture and/or pain preventing shoulder elevation above 90 degrees.
* Body mass index > 30 kg/m2 (severe obesity)
* Known abdominal or aortic aneurysm
* Known atrial of ventricular arrhythmia, unstable hypertension,
* Diabetes with a history of recurrent hypoglycemic episodes
* Cognitive impairments, such as co-morbid brain injury, depression, and/or mental illness preventing an active participation in the study
* Known contact allergy to silver
* Grade three pressure sore or cellulitis in the region intended to be tested
* Body jewelry or tattoos in the area to be stimulated (between sites of the electrodes and/or at less than 2 inch distance from electrodes).

Specifically for participants with SCI:

* Recurrent episodes of orthostatic hypotension preventing a prolonged seated position, or recurrent uncontrolled autonomic dysreflexia episodes
* Prior history of myocardial infarction or stroke

Specifically for participants with Stroke:

* Hemianopia, body hemineglect and/or aphasia preventing an efficient communication with researcher and interaction with the garment and the objects.
* Prior history of spinal cord injury

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Wolf Motor Function Test | Baseline
  For participants who had a stroke. A series of movement and object manipulations video-taped, timed, and rated for their quality of execution and success.
  The TRI-Hand Function Test is a gross motor function test used to assess upper extremity function in SCI. There are two components of the test an object manipulation component and a strength measurement component.
  The Wolf Motor Function Test is validated in stroke and it consists of performing 17 tasks (moving the hand on certain spots, handling daily life objects). The evaluator scores the quality of movement (e.g. 0 = does not attempt; 3. = movement with synergy, effort, at low speed; 5 = movement appears to be normal).
Toronto Rehabilitation Institute Hand Function Test | Baseline
  For participants who had a spinal cord injury. A series of movement and object manipulations video-taped, timed, and rated for their quality of execution and success.
Wolf Motor Function Test | End study, after 14 weeks on average
  For participants who had a stroke. A series of movement and object manipulations video-taped, timed, and rated for their quality of execution and success.
  Re-measured after the participant completed the 40 sessions
Toronto Rehabilitation Institute Hand Function Test | End study, after 14 weeks on average
  For participants who had a spinal cord injury. A series of movement and object manipulations video-taped, timed, and rated for their quality of execution and success.
  Re-measured after the participant completed the 40 sessions

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) | Baseline
  The FIM is a 12 item ordinal scale used to assess progress during rehabilitation and measures independent performance in various domains of activities of daily living.
  FIM score ranges from 12 to 84 FIM will be administered only in participants with Stroke.
Functional Independence Measure (FIM) | End study, after 14 weeks on average
  The FIM is a 12 item ordinal scale used to assess progress during rehabilitation and measures independent performance in various domains of activities of daily living.
  FIM score ranges from 12 to 84 FIM will be administered only in participants with Stroke. Re-measured after the participant completed the 40 sessions
Spinal Cord Independence Measure | Baseline
  SCIM is a disability scale that has been specifically developed to evaluate functional outcomes in patients with SCI. It assess function in three core areas 1. Self care 2.Respiration and 3.Mobility.
  The SCIM scores range from 0 to 100 points. SCIM will be administered only in participants with SCI.
Spinal Cord Independence Measure | End study, after 14 weeks on average
  SCIM is a disability scale that has been specifically developed to evaluate functional outcomes in patients with SCI. It assess function in three core areas 1. Self care 2.Respiration and 3.Mobility.
  The SCIM scores range from 0 to 100 points. SCIM will be administered only in participants with SCI. Re-measured after the participant completed the 40 sessions
Grip strength | Baseline
  Average of the 3 maximal grip strength recorded with a Digital Grip Hand Dynamometer.
  For both group.
Grip strength | End study, after 14 weeks on average
  Average of the 3 maximal grip strength recorded with a Digital Grip Hand Dynamometer. Re-measured after the participant completed the 40 sessions For both group.
Set-up time | During the procedure
  Record with a stop watch the time required to 1. put on the FES-garment, 2. wet the electrodes, and 3. select the appropriate stimulation intensity.
Execution of the training tasks with FES | During the procedure
  Record in the CRF of the weight of bottle lifted at shoulder level while receiving FES.
Execution of the training tasks without FES | During the procedure
  Record in the case report form (CRF) of the highest weight of bottle lifted at shoulder level without delivery of FES.

CONTACTS AND LOCATIONS:
Overall Officials: Milos R Popovic, PhD, Principal Investigator — Toronto Rehabilitation Institute
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
This aspect hasn't been discussed with all collaborators of the study.

REFERENCES:
- [Background] Zhou H, Lu Y, Chen W, Wu Z, Zou H, Krundel L, Li G. Stimulating the Comfort of Textile Electrodes in Wearable Neuromuscular Electrical Stimulation. Sensors (Basel). 2015 Jul 16;15(7):17241-57. doi: 10.3390/s150717241. PMID 26193273
- [Background] Kapadia NM, Zivanovic V, Furlan JC, Craven BC, McGillivray C, Popovic MR. Functional electrical stimulation therapy for grasping in traumatic incomplete spinal cord injury: randomized control trial. Artif Organs. 2011 Mar;35(3):212-6. doi: 10.1111/j.1525-1594.2011.01216.x. PMID 21401662
- [Background] Kawashima N, Popovic MR, Zivanovic V. Effect of intensive functional electrical stimulation therapy on upper-limb motor recovery after stroke: case study of a patient with chronic stroke. Physiother Can. 2013 Winter;65(1):20-8. doi: 10.3138/ptc.2011-36. PMID 24381377
- [Background] Eraifej J, Clark W, France B, Desando S, Moore D. Effectiveness of upper limb functional electrical stimulation after stroke for the improvement of activities of daily living and motor function: a systematic review and meta-analysis. Syst Rev. 2017 Feb 28;6(1):40. doi: 10.1186/s13643-017-0435-5. PMID 28245858